CLINICAL TRIAL: NCT06272175
Title: Immediate Effects of Open and Closed Kinetic Chain Activities on Upper Extremity Spasticity and Motor Dexterity in Stroke Patients"
Brief Title: Immediate Effects of Open and Closed Kinetic Chain Exercises on Upper Extremity in Stroke Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10102023
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; Spasticity; Dexterity; Open Kinetic Chain; Closed Kinetic Chain
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Kinetic Chain Activity Group (Experimental): Open kinetic chain activity will involve Flexion-Abduction-External Rotation and Flexion-Adduction-External Rotation patterns from the Proprioceptive Neuromuscular Facilitation (PNF). During the application, participants will lie on their back, and the pattern will be initiated from the opposite direction of the targeted movement. Participants will be encouraged to perform the movement as actively as possible. Assistance will be provided if the participant cannot complete the pattern. No other PNF techniques will be applied. Both patterns will be practiced for 10 repetitions. Resting periods will be provided as needed to prevent fatigue. The entire application is planned to last approximately 5 minutes.
  Interventions: Other: Open Kinetic Chain Activity
- Closed Kinetic Chain Activity Group (Experimental): For closed kinetic chain activity of the upper extremity, an activity involving weight shifting onto the hands on a table while standing with the elbows in extension will be used. Participants will be asked to shift weight onto the hemiplegic upper extremity for 30 seconds. After a 30-second rest period, the weight shifting will be repeated for a second time.
  Interventions: Other: Closed Kinetic Chain Activity

INTERVENTIONS:
Other: Open Kinetic Chain Activity — PNF Flexion-Abduction-External Rotation and Flexion-Adduction-External Rotation patterns will be actively performed on the hemiplegic upper extremity.
  Arms: Open Kinetic Chain Activity Group
Other: Closed Kinetic Chain Activity — Weight-bearing on the hemiplegic hand with extended elbow in standing position
  Arms: Closed Kinetic Chain Activity Group

SUMMARY:
Stroke is a sudden disruption of blood flow to the brain, resulting in physical and mental disabilities. It's a global health issue affecting millions each year, often leading to paralysis, altered muscle tone, and loss of motor control and balance. This study aims to examine the immediate effects of open and closed kinetic chain activites on upper extremity spasticity and motor dexterity in hemiplegic patients. This study will be conducted simultaneously at İstinye University Hospital Medical Park Gaziosmanpaşa and İstinye University Physiotherapy and Rehabilitation Application and Research Center (İSÜFİZYOTEM). 50 stroke patients will be included in the study, and all participants will be asked to sign an informed consent form. At the beginning of the session, all participants will be evaluated for their socio-demographic characteristics by a questionnaire created by the researchers, muscle viscoelastic properties by MyotonPRO, upper extremity muscle tone by Modified Ashworth Scale, upper extremity motor dexterity by Box and Block Test, and upper extremity joint range of motion by goniometer and by a phone application named as PhysioMaster. After the assessment, participants will be randomly assigned to two groups: open kinetic chain activity group and closed kinetic chain activity group. After performing the exercises, all evaluations will be conducted again. Thus, the aim is to understand the immediate effects of two different group exercises on the evaluated parameters.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis;
* Hemiplegia;
* Subacute&chronic phase (more than 3 months);
* Brunnstrom 3-4-5;
* Unsupported sitting ability;
* Being volunteer.

Exclusion Criteria:

* Having Botox within the last 6 months;
* 4 according to Modified Ashworth Scale;
* Other neurological diagnosis other than stroke.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
MyotonPRO digital palpation device | 6 minutes
  This device is a patented, certified, digital measurement device that measures the amount of tissue displacement that occurs per unit force applied by a probe pressed perpendicularly to the skin overlying the muscle. It measures the viscoelastic properties of the muscles. Latissimus Dorsi will be measured from a point 5 cm above the lower corner of the scapula with the shoulder in 80 flexion. Pectoralis Major will be measured three-quarters of the way from the line between the sternum and the nodule prominence. Measurement of the Biceps Brachii and Brachioradialis muscles will be made from the most swollen points of the muscles. For measurement of the Flexor Carpi Radialis muscle, patients will be taken supine, with the forearm supinated and the elbow approximately 40 degrees flexed, at the one-third (approximately) point of the distance between the elbow line and the lateral side of the ulnar styloid. All measurements will be repeated 3 times and the average will be calculated.
Box and Block Test | 1 minute
  It is a standardized assessment used to measure upper extremity motor dexterity. It involves moving blocks from one side of a box to the other within a minute. It is a clinic-friendly standardized assessment that is portable, easy to obtain, simple to administer, and can be administered quickly without a specific setting.

SECONDARY OUTCOMES:
Modified Ashworth Scale | 3 minutes
  Upper extremity spasticity level of participants will be evaluated with the Modified Ashworth Scale (MAS). In the MAS evaluation, participants were in a supine position, with the arms next to the body and the shoulder in slight abduction. Shoulder adductors, elbow flexors and wrist flexors will be assessed.
Goniometer | 5 minutes
  It will be used to measure the range of motion. Shoulder flexion and abduction, elbow extension, supination and pronation, and wrist extension, ulnar & radial deviation will be measured.
PhysioMaster | 5 minutes
  This phone application will be used to measure the range of motion. Shoulder flexion and abduction, elbow extension, supination and pronation, and wrist extension, ulnar & radial deviation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Can, Study Chair — Istinye University; Seyhan Söyüncü, Study Chair — Istinye University
Locations (1):
- Istinye University Hospital Medical Park Gaziosmanpasa, Istanbul, Turkey (Türkiye)